CLINICAL TRIAL: NCT00508599
Title: Effect of a 2-day Bed Rest on Metabolic and Cardiovascular Risk Factors in Type 2 Diabetic Patients
Brief Title: The Effects of Two Days of Bedrest on Insulin Resistance in Type 2 Diabetics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Responsible Party: David S. Schade, M.D., University of New Mexico
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 03-163
Record Dates: First submitted 2007-07-26; First posted 2007-07-30 (Estimated); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Type 2 Diabetes; Insulin Resistance
Keywords: type 2 diabetes; bed rest; insulin resistance; insulin; glucose; orthostatic response
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (No Intervention): Study 1 is the control arm in which participants continue with their normal activity.
- 2. (Experimental): Study 2 consists of 48 hours of complete bed rest.
  Interventions: Other: Study 2 (48 hours of complete bed rest)

INTERVENTIONS:
Other: Study 2 (48 hours of complete bed rest) — Effects of 48 hours of bed rest on insulin resistance in type 2 diabetic subjects.
  Arms: 2.

SUMMARY:
The hypothesis of this study is that bed rest in diabetic patients will result in a deterioration of metabolic control (primarily glucose).

Specific aims:

1. To determine the change in metabolic control in type 2 diabetic individuals when three days of bed rest is compared to three days of activity;
2. To determine the rate of progression of the deterioration in metabolic control and the magnitude of the decrease;
3. To assess whether the anticipated deterioration of metabolic control has effects on several parameters of glucose metabolism, including hyperglycemia and hypoglycemia;
4. To determine the effects of bed rest on surrogate markers of atherosclerosis, such as plasminogen activator inhibitor 1 (PAI1), C-reactive protein (CRP), and homocysteine.
5. To compare the effects of 48 hours of bed rest on orthostatic responses in type 2 diabetic patients, and healthy non-diabetics.
6. To make recommendations to the diabetic community to prevent metabolic deterioration during a 3 day hospitalization.

DETAILED DESCRIPTION:
The goal for all diabetic patients is to maintain their metabolic control as close to normal as possible to prevent the short and long term complications of diabetes. Surgery of any type presents a unique challenge to the diabetic patient because two factors tend to worsen their metabolic control 1) the stress of the actual surgery and 2) the bed rest that follows the surgery. Data has clearly shown that surgery increase counter regulatory hormones (epinephrine, glucagon, growth hormone and cortisol). What has not been studied is the effect of bed rest per se on metabolic control. This is surprising because there are many studies in normal healthy people demonstrating that simple bed rest increases insulin resistance and worsens metabolic control.

The proposed study will define the metabolic effects of simple, three-day bed rest on metabolic control in healthy type 2 diabetic volunteers while evaluating the orthostatic response after bed rest. All studies will be done in the inpatient, General Clinical Research Center (GCRC). All volunteers will stop their oral antidiabetic medication before they enter the GCRC. They will be placed on intravenous insulin to prevent severe metabolic deterioration and hyperglycemia. The amount of insulin we have to give them to maintain metabolic control will be one measure of the effects of bed rest on metabolic control.

Experimental Design and Methods.

A crossover study in twenty healthy normal and twenty healthy type 2 diabetic subjects will be utilized. Each subject will be admitted the the GCRC the night prior to beginning the study in order to insure metabolic stability at the start of the protocol. Each subject will stay in the GCRC three full days (three nights) from the time of admission. Each subject will be admitted on two separate occasions, separated by at least a two week interval. A diagram of the protocol is given below:

The primary difference between the two admissions will be the amount of physical activity allowed each subject. On the normal physical activity GCRC admission, the subject will be encouraged to stay our of bed until his/her usual bedtime. All procedures and meals will take place in the GCRC but in between times the subject will be encouraged to walk around the hospital and to carry out normal activities of daily living. On the bed rest GCRC admission, the subjects will be encouraged to stay in bed as much as possible and to use a bedside commode. A tilt test was performed on the morning of the first day of each hospitalization and again 48 hours later. The same testing will be done as in the normal activity admission.

All medications that the volunteer usually takes at home will be continued in the hospital.

The volunteer will be in the GCRC for three days: Day 1, Day 2, and Day 3. The following tests will be done on the three days:

Day 1 - Blood will drawn for fasting lipids, glucose, insulin, and C-peptide as well as surrogate markers of atherosclerosis including PAI-1, IL-6, homocysteine, fibrinogen, and CRP. In addition, a tilt table test will be done to assess autonomic response to activity or bedrest.

Day 2 - Blood will drawn for fasting lipids, glucose, insulin, and C-peptide as well as surrogate markers of atherosclerosis including PAI-1, IL-6, homocysteine, fibrinogen, and CRP.

Day 3 - Blood will drawn for fasting lipids, glucose, insulin, and C-peptide as well as surrogate markers of atherosclerosis including PAI-1, IL-6, homocysteine, fibrinogen, and CRP. In addition, a tilt table test will be done to assess autonomic response to activity or bed rest.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetic for at least 6 months.
* Healthy volunteers.
* Type 2 diabetic subjects will have some nominal ability to secrete endogenous insulin as demonstrated by a post-stimulation C-peptide concentration of at least 6 ng/ml.
* All subjects will be mentally fit to give informed consent.
* Hemoglobin A1C value below 11% (normal range = 4.4-5.8%) prior to study enrollment.

Exclusion Criteria:

* Hemoglobin A1c values > 11%
* Severe cardiovascular, hepatic, or renal disease
* Past current history of drug or alcohol abuse
* Diabetic gastroparesis
* Uncontrolled hypertension ( > 140-90 mmHg)
* Marked hyperlipidemia (serum LDL > 158mg/dl, or serum TG >691 mg/dl)
* Medications that interfere with glucose homeostasis
* Coumadin or other anticoagulation medications
* History of thrombosis or thrombophlebitis
* Current malignancy
* Smoker
* Pregnancy
* Contact precautions

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2003-01 (Actual); Primary Completion 2004-01 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Insulin resistance and orthostatic response | 48 hours bed rest and 48 hours activity

SECONDARY OUTCOMES:
Change in glucose, insulin, and orthostatic impairment. | 48 hours of bed rest and 48 hours of Activity

CONTACTS AND LOCATIONS:
Overall Officials: David S Schade, M.D., Principal Investigator — University of New Mexico
Locations (1):
- University of New Mexico, Clinical Translational Science Center, Albuquerque, New Mexico, United States

REFERENCES:
- [Background] Smorawinski J, Kaciuba-Uscilko H, Nazar K, Kubala P, Kaminska E, Ziemba AW, Adrian J, Greenleaf JE. Effects of three-day bed rest on metabolic, hormonal and circulatory responses to an oral glucose load in endurance or strength trained athletes and untrained subjects. J Physiol Pharmacol. 2000 Jun;51(2):279-89. PMID 10898100
- [Background] Nichiporuk IA, Evdokimov VV, Erasova VI, Smirnov OA, Goncharova AG, Vassilieva GYu, Vorobiev DV. Male reproductive system in conditions of bed-rest in a head-down tilt. J Gravit Physiol. 1998 Jul;5(1):P101-2. PMID 11542307
- [Background] Stuart CA, Shangraw RE, Prince MJ, Peters EJ, Wolfe RR. Bed-rest-induced insulin resistance occurs primarily in muscle. Metabolism. 1988 Aug;37(8):802-6. doi: 10.1016/0026-0495(88)90018-2. PMID 3043146
- [Background] Yanagibori R, Suzuki Y, Kawakubo K, Makita Y, Gunji A. Carbohydrate and lipid metabolism after 20 days of bed rest. Acta Physiol Scand Suppl. 1994;616:51-7. PMID 8042526
- [Background] Blanc S, Normand S, Pachiaudi C, Fortrat JO, Laville M, Gharib C. Fuel homeostasis during physical inactivity induced by bed rest. J Clin Endocrinol Metab. 2000 Jun;85(6):2223-33. doi: 10.1210/jcem.85.6.6617. PMID 10852455
- [Background] Mikines KJ, Richter EA, Dela F, Galbo H. Seven days of bed rest decrease insulin action on glucose uptake in leg and whole body. J Appl Physiol (1985). 1991 Mar;70(3):1245-54. doi: 10.1152/jappl.1991.70.3.1245. PMID 2032990
- [Background] Yanagibori R, Kondo K, Suzuki Y, Kawakubo K, Iwamoto T, Itakura H, Gunji A. Effect of 20 days' bed rest on the reverse cholesterol transport system in healthy young subjects. J Intern Med. 1998 Apr;243(4):307-12. doi: 10.1046/j.1365-2796.1998.00303.x. PMID 9627145
- [Background] Valek J, Valkova L, Vlasakova Z, Topinka V. Increased fibrinogen levels in the offspring of hypertensive men. Relation with hyperinsulinemia and the metabolic syndrome. Arterioscler Thromb Vasc Biol. 1995 Dec;15(12):2229-33. doi: 10.1161/01.atv.15.12.2229. PMID 7489247
- [Background] Gough SC, Rice PJ, McCormack L, Chapman C, Grant PJ. The relationship between plasminogen activator inhibitor-1 and insulin resistance in newly diagnosed type 2 diabetes mellitus. Diabet Med. 1993 Aug-Sep;10(7):638-42. doi: 10.1111/j.1464-5491.1993.tb00137.x. PMID 8403825
- [Derived] Schneider SM, Robergs RA, Amorim FT, de Serna DG, Duran-Valdez EE, Schade DS. Impaired orthostatic response in patients with type 2 diabetes mellitus after 48 hours of bed rest. Endocr Pract. 2009 Mar;15(2):104-10. doi: 10.4158/EP.15.2.104. PMID 19289319
- [Derived] Duran-Valdez E, de Serna DG, Schneider S, Amorim F, Burge M, Schade DS. Metabolic effects of 2 days of strict bed rest. Endocr Pract. 2008 Jul-Aug;14(5):564-9. doi: 10.4158/EP.14.5.564. PMID 18753098